CLINICAL TRIAL: NCT02409979
Title: Impact of Carbon Dioxide Insufflation and Water Exchange on Post-Colonoscopy Outcomes: A Randomized Controlled Trial
Brief Title: Impact of Carbon Dioxide Insufflation and Water Exchange on Post-Colonoscopy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Ospedaliero Santa Barbara (Other)
Responsible Party: Principal Investigator, Sergio Cadoni, M.D., Responsabile Servizio Endoscopia Digestiva, Presidio Ospedaliero Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PG.2015/3645; Delibera 387/C 17 Marzo 2015 (Other: Azienda USL 07 Carbonia, Regione Sardegna)
Record Dates: First submitted 2015-03-23; First posted 2015-04-07 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Abdominal Pain
Keywords: colonoscopy; carbon dioxide; water exchange; discomfort; colonoscopy pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Carbon dioxide method (Active Comparator): Colonoscopy performed as usual, with the minimal CO2 insufflation required to aid insertion and adequate distension during withdrawal for exploration. Washing allowed as needed. Considered to be standard procedure.
  Interventions: Other: Carbon dioxide method
- Water Exchange-CO2 (Experimental): Insufflation not used until the cecum is reached. Infusion of a sufficient amount of water to render the lumen a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for opaque water. Air pockets and residual feces will be always aspirated. Withdrawal phase done using carbon dioxide insufflation.
  Interventions: Other: Water Exchange-CO2
- Water Exchange-AI (Experimental): Insufflation not used until the cecum is reached. Infusion of a sufficient amount of water to render the lumen a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for opaque water. Air pockets and residual feces will be always aspirated. Withdrawal phase done using air insufflation.
  Interventions: Other: Water Exchange-AI

INTERVENTIONS:
Other: Carbon dioxide method — Insufflation with CO2 during insertion and withdrawal phases of colonoscopy.
  Arms: Carbon dioxide method
Other: Water Exchange-CO2 — Insertion using water exchange, withdrawal using CO2 insufflation.
  Arms: Water Exchange-CO2
Other: Water Exchange-AI — Insertion using water exchange, withdrawal using air insufflation.
  Arms: Water Exchange-AI

SUMMARY:
Room air insufflated during colonoscopy cannot be completely suctioned, is not easily absorbed and remains in the bowel for quite some time, resulting in prolonged bowel distension with the discomfort of bloating. Sufferers often experience a sensation of fullness and abdominal pressure, relieved only after expulsion of the residual gas, often accompanied by colic pain. This can be a lengthy process, and some patients continue to report pain as long as 24 hours after the procedure. Abdominal discomfort after colonoscopy is an adverse event commonly reported by patients, and definitely associated with the procedure. Published reports show that the use of carbon dioxide (CO2) insufflation significantly decreases bloating and pain up to 24 hours post-procedure. Preliminary results of the investigators' previous study about on-demand sedation colonoscopy in diagnostic patients showed that, compared with CO2 insufflation, the water exchange group (WE, infusion of water to distend the lumen during insertion; suction of infused water, residual air pockets an feces predominantly during insertion) achieved significantly lower real-time insertion pain scores. Moreover (insertion-withdrawal method) WE-CO2 had the lowest bloating scores just after the procedure and at discharge, comparable with those achieved by CO2-CO2. Compared with WE-CO2, the use of WE-air insufflation (AI) showed significantly higher bloating scores just after the procedure and at discharge; compared with CO2-CO2 differences were significant only at discharge. The investigators decided to conduct a prospective randomized controlled trial comparing WE-CO2, WE-AI and CO2-CO2. The investigators will test the hypothesis that patients examined by the combination of WE-CO2 will have significantly lower bloating scores at specific time points after colonoscopy than those examined using WE-AI or CO2-CO2. The investigators will also assess the impact of these three methods on patients comfort and activities in the post-procedure period.

DETAILED DESCRIPTION:
Design: Prospective double blinded two-center randomized controlled trial. Methods: Colonoscopy with CO2 insufflation and water exchange-CO2, water exchange-AI; split-dose bowel preparation; on demand-sedation.

Control method: CO2 insufflation colonoscopy. Study methods: water exchange-CO2 colonoscopy, water exchange-AI colonoscopy.

Population: Consecutive 18 to 80 year-old first-time diagnostic outpatients. After informed consent, assignment to control or study arms based on computer generated randomization list with block allocation and stratification.

ELIGIBILITY:
Inclusion Criteria:

* consecutive 18 to 80 year-old first-time diagnostic outpatients agreeing to start procedure without premedication

Exclusion Criteria:

* patient unwillingness to start the procedure without sedation/analgesia
* previous colorectal surgery
* proctosigmoidoscopy or bidirectional endoscopy
* patient refusal or inability to provide informed consent
* inadequate consumption of bowel preparation
* moderate or severe chronic obstructive pulmonary disease requiring oxygen
* medical history of CO2 retention
* history of inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in abdominal bloating sensation after colonoscopy. | Within the first 24 hours after the procedure.
  Change of patients' sensation of abdominal bloating. Assessed by blinded observer just after examination, at discharge; and at 1, 3, 6, 12 and 24 hours after the procedure using a questionnaire given to patients. Measured on an eleven-point Numeric Rating Scale (NRS): 0=none, 10=full bloating. Results will be recorded by telephone recall.

SECONDARY OUTCOMES:
Change in pain score after colonoscopy. | Within the first 24 hours after the procedure.
  Assessed by blinded observer just after examination, at discharge; and at 1, 3, 6, 12 and 24 hours after the procedure using a questionnaire given to patients. Measured using an eleven-point NRS (0=none, 10=maximum pain). Results will be recorded by telephone recall.
Real-time insertion pain. | 1 hour.
  Pain assessed using a NRS (0=absence of pain, 2=simply "discomfort", 10=worst pain). Before the procedure, an endoscopic nurse will explain the NRS scoring system to the patients. At irregular intervals during colonoscopy (around 60 seconds) assisting nurse will ask patients about discomfort or pain. The responses will be recorded, and the maximum pain score noted. Colonoscopists not participating in gathering the informations.
Number of episodes of incontinence or of soiled underwear experienced in the 6 hours after colonoscopy. | 6 hours.
  Recorded at discharge and assessed post-procedure up to 6 hours using a questionnaire given to patients. Results will be recorded by telephone recall.
Number of flatus episodes post-procedure. | 24 hours.
  Recorded at discharge and assessed post-procedure up to 24 hours using a questionnaire given to patients. Results will be recorded by telephone recall.
Number of incontinence episodes post-procedure. | 6 hours.
  Recorded at discharge and assessed post-procedure up to 6 hours using a questionnaire given to patients. Results will be recorded by telephone recall.
Toilet use for bowel movement post-procedure. | 6 hours.
  Recorded at discharge and assessed post-procedure up to 6 hours using a questionnaire given to patients. Results will be recorded by telephone recall.
Patients' satisfaction with the procedure. | 24 hours.
  Assessed post-procedure after 24 hours using a questionnaire given to patients (0=not satisfied, 10=very satisfied). Results will be recorded by telephone recall.
Willingness to repeat colonoscopy. | 24 hours.
  Assessed post-procedure after 24 hours using a questionnaire given to patients (0=not willing to repeat, 10=very likely to repeat). Results will be recorded by telephone recall.
Interference of colonoscopy on work/normal activities the same day of the procedure. | Up to 12 hours.
  Assessed post-procedure after 12 hours using a questionnaire given to patients (0=nothing at all, 10=a lot). Results will be recorded by telephone recall.
Day of work missed the day after the procedure. | 24 hours.
  Work activities missed the day after colonoscopy due to some effect of the procedure (yes, no). Assessed post-procedure after 24 hours using a questionnaire given to patients. Results will be recorded by telephone recall.

OTHER OUTCOMES:
Cecal intubation rate. | 1 hour.
  Cecal intubation will be defined as reaching beyond the ileocecal valve with adequate visualization of the appendix orifice.
Cecal intubation time. | 1 hour.
  Defined as the time for passage of the colonoscope from the rectum to the cecum.
Total procedure time. | 1 hour.
  Total procedure time (including time required for water infusion, polyp resection or biopsy).
Adenoma detection rate. | 9 months.
  Proportion of subjects with at least one adenoma of any size.
On-demand sedation. | 1 hour.
  Offered at patient request for a NRS score ≥2. Medications given as per institutional regulation. Dose titrated based on patients' reported real-time pain score, age, weight and comorbidity.
Oxygen desaturation. | 1 hour.
  Significant oxygen desaturation (<85% for >15 seconds) will be recorded.
Vagal reaction. | 1 hour.
  Vagal reaction (heart rate <60 beats per minute accompanied by excessive sweating, nausea and/or vomiting) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cadoni, MD, Principal Investigator — S. Barbara Hospital, Iglesias (CI) Italy
Locations (3):
- Sepulveda Ambulatory Care Center, VA Greater Los Angeles Healthcare System, Los Angeles, California, United States
- Digestive Diseases Center, Vìtkovice Hospital, Ostrava, Czechia
- Digestive Endoscopy Unit, Ospedale S. Barbara, Iglesias, CI, Italy

REFERENCES:
- [Result] Sumanac K, Zealley I, Fox BM, Rawlinson J, Salena B, Marshall JK, Stevenson GW, Hunt RH. Minimizing postcolonoscopy abdominal pain by using CO(2) insufflation: a prospective, randomized, double blind, controlled trial evaluating a new commercially available CO(2) delivery system. Gastrointest Endosc. 2002 Aug;56(2):190-4. doi: 10.1016/s0016-5107(02)70176-4. PMID 12145595
- [Result] Zubarik R, Fleischer DE, Mastropietro C, Lopez J, Carroll J, Benjamin S, Eisen G. Prospective analysis of complications 30 days after outpatient colonoscopy. Gastrointest Endosc. 1999 Sep;50(3):322-8. doi: 10.1053/ge.1999.v50.97111. PMID 10462650
- [Result] de Jonge V, Sint Nicolaas J, van Baalen O, Brouwer JT, Stolk MF, Tang TJ, van Tilburg AJ, van Leerdam ME, Kuipers EJ; SCoPE consortium. The incidence of 30-day adverse events after colonoscopy among outpatients in the Netherlands. Am J Gastroenterol. 2012 Jun;107(6):878-84. doi: 10.1038/ajg.2012.40. Epub 2012 Mar 6. PMID 22391645
- [Result] Lee YC, Wang HP, Chiu HM, Lin CP, Huang SP, Lai YP, Wu MS, Chen MF, Lin JT. Factors determining post-colonoscopy abdominal pain: prospective study of screening colonoscopy in 1000 subjects. J Gastroenterol Hepatol. 2006 Oct;21(10):1575-80. doi: 10.1111/j.1440-1746.2006.04145.x. PMID 16928219
- [Result] Falt P, Liberda M, Smajstrla V, Kliment M, Bartkova A, Tvrdik J, Fojtik P, Urban O. Combination of water immersion and carbon dioxide insufflation for minimal sedation colonoscopy: a prospective, randomized, single-center trial. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):971-7. doi: 10.1097/MEG.0b013e3283543f16. PMID 22569079
- [Derived] Cadoni S, Falt P, Gallittu P, Liggi M, Smajstrla V, Leung FW. Impact of carbon dioxide insufflation and water exchange on postcolonoscopy outcomes in patients receiving on-demand sedation: a randomized controlled trial. Gastrointest Endosc. 2017 Jan;85(1):210-218.e1. doi: 10.1016/j.gie.2016.05.021. Epub 2016 May 17. PMID 27207825